Study ID:IRB201601774 Date Approved: 10/18/2017 Expiration Date: 11/2/2018

NCT02930824






| INFORMED CONSENT FORM to Participate in Research, and |
|---|
| AUTHORIZATION<br>to Collect, Use, and Disclose Protected<br>Health Information (PHI) |
| INTRODUCTION |
| Name of person seeking your consent: |

Please read this form, which describes the study in some detail. A member of the research team will describe this study to you and answer all of your questions. Your participation is entirely voluntary. If you choose to participate you can change your mind at any time and withdraw from the study. You will not be penalized in any way or lose any benefits to which you would otherwise be entitled if you choose not to participate in this study or to withdraw. If you have questions about your rights as a research subject, please call the University of Florida Institutional Review Board (IRB) office at (352) 273-9600.

Place of employment & position:

### **GENERAL INFORMATION BOUT THIS STUDY**

1. Name of Participant ("Study Subject")

\_\_\_\_\_\_

2. What is the Title of this research study?

Implementing Genomics in Practice (IGNITE) Proof of Concept Study: CYP2C19 genotype-supported versus conventional Proton Pump Inhibitor dosing

3. Who do you call if you have questions about this research study?

Principal Investigator: Larisa Cavallari, Pharm.D., Phone: 352-273-8245

IRB Project #: 201601774 IRB Version: 10/19/2011



#### 4. Who is paying for this research study?

The sponsor of this study is the National Institutes of Health (NIH).

#### 5. Why is this research study being done?

The purpose of this research study is to find out if information about an individual's genetic makeup (DNA) will help doctors improve the treatment of gastroesophagel reflux disease, commonly called heartburn, or symptoms of indigestion. Symptoms may include sharp or burning pain in your chest, tightness in your chest or upper abdomen, stomach cramps, nausea, hoarseness, sore throat, coughing, sour or bitter taste in your mouth, and trouble swallowing. Genetic makeup is what determines a person's body traits, such as eye color and height. It also may determine how quickly or slowly your body removes medication from your system. People's body traits differ from one another because genetic makeup differs from person to person. By participating in this study, investigators can find out if your genes can help doctors choose better medication doses to decrease symptoms of heartburn or indigestion. This will be done through surveys to be completed by you at the beginning and end of your participation. Through this study, we will also be able to gain a better understanding of how this genetic testing can inform your doctor's decisions for your treatment.

You are being asked to be in this research study because your doctor has prescribed a medication for you called a proton pump inhibitor to help decrease your symptoms of heartburn or indigestion.

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

### WHAT CAN YOU EXPECT IF YOU PARTICIPATE IN THIS STUDY?

# 6. What will be done as part of your normal clinical care (even if you did not participate in this research study)?

You will continue to receive the same clinical care your doctor is currently providing to help manage your heartburn or symptoms of indigestion.

### 7. What will be done only because you are in this research study?

If you choose to participate in this study a blood sample will be collected from you. A trained and qualified member of our study staff or phlebotomist will draw your blood by putting a needle into a vein in your arm. About 1 teaspoonful of blood will be taken. This blood will be used to assess your specific genetic profile within 1 gene to

IRB Project #: 201601774 



help your doctor determine the best treatment plan for your heartburn or symptoms of indigestion.

You will be randomly assigned (like the flip of a coin) into either the test group or the control group, and there is a 50-50 chance that will be in either group. Research studies of this type usually compare a "test" group and a "control" group when trying to determine if information gained from genetic makeup is helpful to doctors in making decisions about what medication to prescribe to patients. Regardless of which group you are randomly assigned to, your blood sample will be sent to the UF Health laboratory, and your genetic makeup will be determined using your blood.

You will find out which group you have been assigned to at your next visit with your doctor. If you are assigned to the test group, your genetic test results will be shared with your doctor and placed in your medical record in about 2 weeks to help support your doctor's decision in treatment selection for your heartburn or symptoms of indigestion. If you are assigned to the control group, your genetic test results will not be available to your doctor until the end of your participation in this study, and selection of your medication and treatment plan will be made by your doctor based upon his/her best clinical judgment only. In the future, your doctor can use the information from the genetic test to help support your treatment for heartburn or indigestion, if we find out that this information helps.

You will be asked to complete three short surveys at the beginning of the study and again as close to 3 months after the first survey as possible for research purposes. The surveys at 3 months can be completed during your regularly scheduled visit with your physician or by telephone if you do not have an appointment scheduled in 3 months. The first two questionnaires are about your heartburn or indigestion symptoms. Your doctor and other researchers will use this information to compare how well your heartburn or indigestion symptoms were controlled before and after the study. We will compare how well heartburn relief and/or indigestion symptoms were controlled in patients who had their genetic information used for managing their symptoms and those who did not have this information used. A third questionnaire will ask you what you know and how you feel about genetic testing to help with drug prescribing. These surveys should take 15 to 20 minutes to complete.

Researchers for the study will look at your medical record for information about your health and medications in the 24 months after you are enrolled in the study.

Medical data about you will be collected during your participation in this study. After the study is completed your name and any other identifiable information is removed, your data will no longer be able to be linked to you. At the end of this form you will be given the choice to not have your data stored for future unknown research.

De-identified datasets may be shared with the other site investigators of the sponsor listed in question 4 to be used for network wide analysis.

If you have any questions now or at any time during the study, please contact one of the research team members listed in question 3 of this form.

IRB Project #: 201601774 
IRB Version: 10/19/2011



#### 8. How long will you be in this research study?

Your active participation in this study will last until the completion of the final follow up surveys, or about 12 weeks from the time you have your blood drawn. Researchers for this study will also look at your medical record to collect information about your health and medications prescribed during in the 24 months after you enrolled in the study.

#### 9. How many people are expected to take part in this research study?

This study will enroll a total of 200 subjects:120 adult patients like yourself at UF Health and 60 pediatric patients at Nemours Children's Hospital who will participate in this research study. We may also enroll an additional 20 subjects in case some subjects discontinue participation prematurely.

# WHAT ARE THE RISKS AND BENEFITS OF THIS STUDY AND WHAT ARE YOUR OPTIONS?

# 10. What are the possible discomforts and risks from taking part in this research study?

The risks of drawing blood from a vein include discomfort at the site of puncture; possible bruising and swelling around the puncture site; rarely an infection; and, uncommonly, faintness from the procedure. There is a chance that treatment decisions made based on your genetic information could lead to worsening or your symptoms or increased side effects.

A Federal law, called the Genetic Information Nondiscrimination Act (GINA), makes it illegal for health insurance companies, group health plans, and most employers to discriminate against you based on your genetic information. Additional information can be obtained at: http://irb.ufl.edu/gina.html or call 1-800-669-3362. If you think this law has been violated, it will be up to you to pursue any compensation from the offending insurance company and/or employer.

Researchers will take appropriate steps to protect any information they collect about you. However, there is a slight risk that information about you could be revealed inappropriately or accidentally. Depending on the nature of the information, such a release could upset or embarrass you, or possibly affect your insurability or employability. Questions 17-21 in this form discuss what information about you will be collected, used, protected, and shared.

This study may include risks that are unknown at this time.

Participation in more than one research study or project may further increase the risks to you. If you are already enrolled in another research study, please inform one of the

IRB Project #: 201601774 



research team members listed in question 3 of this form or the person reviewing this consent with you before enrolling in this or any other research study or project.

Throughout the study, the researchers will notify you of any new information that may become available and might affect your decision to remain in the study.

If you wish to discuss the information above or any discomforts you may experience, please ask questions now or call one of the research team members listed in question 3 of this form.

#### 11a. What are the potential benefits to you for taking part in this research study?

The genetic test results that are provided as part of this study may be helpful to help your doctor select your treatment for heart burn or indigestion, and in your future medical care, for example, for decisions about the best medications to use if you ever have heart angioplasty done.

#### 11b. How could others possibly benefit from this study?

Other patients who experience heartburn or indigestion may one day have better management due in part to the knowledge gained from the results of this study.

#### 11c. How could the researchers benefit from this study?

In general, presenting research results helps the career of a scientist. Therefore, the Principal Investigator listed in question 3 of this form may benefit if the results of this study are presented at scientific meetings or in scientific journals.

#### 12. What other choices do you have if you do not want to be in this study?

If you choose not to participate in this study, your doctor will choose the medication and treatment plan that he\she feels is appropriate for you. Also since these genetic tests can be ordered by your doctor clinically, this test could be ordered by your doctor outside the study to guide your treatment.

#### 13a. Can you withdraw from this study?

You are free to withdraw your consent and to stop participating in this study at any time. If you do withdraw your consent, you will not be penalized in any way and you will not lose any benefits to which you are entitled. If you decide to withdraw your consent to participate in this study for any reason, please contact one of the research team members listed in question 3 of this form. They will tell you how to stop your participation safely.

If you have any questions regarding your rights as a research subject, please call the Institutional Review Board (IRB) office at (352) 273-9600.

IRB Project #: 201601774 
IRB Version: 10/19/2011



#### 13b. If you withdraw, can information about you still be used and/or collected?

If you discontinue participation in the study (withdraw), the information about you collected up until the time you withdraw can still be used and stored in the data repository in accordance with your choice.

#### 13c. Can the Principal Investigator withdraw you from this study?

You may be withdrawn from the study without your consent for the following reasons:

- At the discretion of the principal investigator or study physician based on what is best for your health and safety.
- If you are a control patient and you or your physician request your genetic test results prior to study completion.

#### WHAT ARE THE FINANCIAL ISSUES IF YOU PARTICIPATE?

#### 14. If you choose to take part in this research study, will it cost you anything?

#### Study Services

The Sponsor will pay for all services required as part of your participation in this study as described above in the question "What Will Be Done Only Because You Are In This Research Study". If you receive a bill for these services, please contact Dr. Larisa Cavallari at (352) 273-8245.

#### Items/Services Not Paid for by the Sponsor

All other medical services provided to you that are not directly required by this study will be billed to you or your insurance company in the usual manner.

#### 15. Will you be paid for taking part in this study?

You will receive a total of \$25 for participating in this study. A \$25 VISA gift card will be provided after your complete your final questionnaire.

If you are in the control group and you or your physician chooses to withdraw your participation to have the genetic information used for clinical care before your study participation is complete, you will receive a \$10 VISA gift card for your study participation up to the point of your withdrawal.

Your payment for participation in this research study is handled through the University of Florida's Human Subject Payment (HSP) Program. Your information which will include your name, address, date of birth, and SSN (depending on amount of money you are paid) is protected. Access to the (HSP) Program site is limited to certain staff with the assigned security role. You will be randomly assigned a specific identification (ID) number to protect your identity.

IRB Project #: 201601774 



The study team will provide you with an informational form called the Prepaid Card Facts document. If you have any problems regarding your payment call the HSP Office (352) 392-9057.

#### 16. What if you are injured because of the study?

If you are injured as a direct result of your participation in this study, only the professional services that you receive from any University of Florida Health Science Center healthcare provider will be provided without charge. These healthcare providers include physicians, physician assistants, nurse practitioners, dentists or psychologists. Any other expenses, including Shands hospital expenses, will be billed to you or your insurance provider.

You will be responsible for any deductible, co-insurance, or co-payments. Some insurance companies may not cover costs associated with research studies or research-related injuries. Please contact your insurance company for additional information.

The Principal Investigator will determine whether your injury is related to your participation in this study.

No additional compensation is routinely offered. The Principal Investigator and others involved in this study may be University of Florida employees. As employees of the University, they are protected under state law, which limits financial recovery for negligence.

Please contact one of the research team members listed in question 3 of this form if you experience an injury or have questions about any discomforts that you experience while participating in this study.

#### 17. How will your health information be collected, used and shared?

If you agree to participate in this study, the Principal Investigator will create, collect, and use private information about you and your health. This information is called protected health information or PHI. In order to do this, the Principal Investigator needs your authorization. The following section describes what PHI will be collected, used and shared, how it will be collected, used, and shared, who will collect, use or share it, who will have access to it, how it will be secured, and what your rights are to revoke this authorization.

Your protected health information may be collected, used, and shared with others to determine if you can participate in the study, and then as part of your participation in the study. This information can be gathered from you or your past, current or future health records, from procedures such as physical examinations, x-rays, blood or urine tests or from other procedures or tests. This information will be created by receiving study treatments or participating in study procedures, or from your study visits and telephone calls. More specifically, the following information may be collected, used, and shared with others:

IRB Project #: 201601774 
IRB Version: 10/19/2011

PI Version: 10/19/2016



- Complete past medical history
- Records of physical exams
- Laboratory and genetic test results
- Results of completed questionnaires
- Medication records
- Clinical outcomes

This information will be stored in locked filing cabinets or on computer servers with secure passwords, or encrypted electronic storage devices.

Some of the information collected could be included in a "limited data set" to be used for other research purposes. If so, the limited data set will only include information that does not directly identify you. For example, the limited data set cannot include your name, address, telephone number, social security number, photographs, or other codes that link you to the information in the limited data set. If limited data sets are created and used, agreements between the parties creating and receiving the limited data set are required in order to protect your identity and confidentiality and privacy.

If you agree to share your genetic information with the National Institutes of Health's database of genotypes and phenotypes (dbGaP) by signing the indicated lines below, the study coordinator will communicate to the laboratory that your de-identified data may be submitted to dbGaP. Your PHI will not be provided to dbGaP, only the result of your genetic test and your non-identifiable demographic information. If you have any questions about what will be shared with dbGaP please ask one of the research study staff listed in question 3 of this form.

### 18. For what study-related purposes will your protected health information be collected, used, and shared with others?

Your PHI may be collected, used, and shared with others to make sure you can participate in the research, through your participation in the research, and to evaluate the results of the research study. More specifically, your PHI may be collected, used, and shared with others for the following study-related purpose(s):

- To determine the effectiveness and side effects of the medications used to help with heartburn relief and/or indigestion symptoms to your genetic information.
- To determine how your survey responses about of the medications used to help with heartburn relief and/or indigestion symptoms are related to your genetic information.

IRB Project #: 201601774 
IRB Version: 10/19/2011



Once this information is collected, it becomes part of the research record for this study.

### 19. Who will be allowed to collect, use, and share your protected health information?

Only certain people have the legal right to collect, use and share your research records, and they will protect the privacy and security of these records to the extent the law allows. These people include:

- The study Principal Investigator and research staff associated with this project.
- Other professionals at the institution where you are participating in the research study.
- the University of Florida Institutional Review Board (IRB; an IRB is a group of people who are responsible for looking after the rights and welfare of people taking part in research) and the University of Florida IRB which is responsible for the approval of this research study.

### 20. Once collected or used, who may your protected health information be shared with?

Your PHI may be shared with:

- The study sponsor (listed in Question 4 of this form).
- United States and agencies who are responsible for overseeing research, such as the Food and Drug Administration, the Department of Health and Human Services, and the Office of Human Research Protections.
- Government agencies who are responsible for overseeing public health concerns such as the Centers for Disease Control and federal, state and local health departments.

Otherwise, your research records will not be released without your permission unless required by law or a court order. It is possible that once this information is shared with authorized persons, it could be shared by the persons or agencies who receive it and it would no longer be protected by the federal medical privacy law.

### 21. If you agree to take part in this research study, how long will your protected health information be used and shared with others?

Your PHI will be used and shared with others until the end of the study, unless you decide to have your information stored in dbGaP. Information stored in dbGaP will be used/shared with others indefinitely.

You are not required to sign this consent and authorization or allow researchers to collect, use and share your PHI. Your refusal to sign will not affect your treatment, payment, enrollment, or eligibility for any benefits outside this research study. However, you cannot participate in this research unless you allow the collection, use

IRB Project #: 201601774 



and sharing of your protected health information by signing this consent and authorization.

You have the right to review and copy your protected health information. However, we can make this available only after the study is finished.

You can revoke your authorization at any time before, during, or after your participation in this study. If you revoke it, no new information will be collected about you. However, information that was already collected may still be used and shared with others if the researchers have relied on it to complete the research. You can revoke your authorization by giving a written request with your signature on it to the Principal Investigator.

IRB Project #: 201601774 IRB Version: 10/19/2011 PI Version: 11/21/2016 Study ID:IRB201601774 Date Approved: 10/18/2017 Expiration Date: 11/2/2018



| SIGNATURES |
|---|
| As an investigator or the investigator's representative, I have explained to the participant the purpose, the procedures, the possible benefits, and the risks of this research study; the alternative to being in the study; and how the participant's protected health information will be collected, used, and shared with others: |
| Signature of Person Obtaining Consent & Authorization Date |
| You have been informed about this study's purpose, procedures, possible benefits, and risks; the alternatives to being in the study; and how your protected health information will be collected, used and shared with others. You have received a copy of this Form. You have been given the opportunity to ask questions before you sign, and you have been told that you can ask questions at any time. |
| You voluntarily agree to participate in this study. You hereby authorize the collection, use and |

sharing of your protected health information as described in sections 17-21 above. By

Date

signing this form, you are not waiving any of your legal rights.

Signature of Person Consenting and Authorizing

IRB Project #: 201601774  IRB Version: 10/19/2011



# Consent to Collect and Store Your Genetic Data for Future Research

As part of the research project the study staff are seeking your consent to store your genetic data.

#### **Reason for Storing Your Data:**

You have recently agreed to participate in the research study listed above, which is funded by the National Institutes of Health (NIH). That research study involves determining certain genetic information about you. The NIH has a policy of sharing genetic information with other researchers to help further new discoveries on disease treatment and cures. Genetic factors are those that people are born with and that can affect other family members. Your genetic information that will be stored in this federal data bank (dbGaP), will be determined by the research study you have already agreed to.

The person in charge of the research project you agreed to (also known as the Principal Investigator) or a representative of the Principal Investigator will describe this data sharing to you and answer all of your questions. Your participation in allowing your data to be shared and stored in this NIH data bank is entirely voluntary. Before you decide whether or not to take part, read the information below and ask questions about anything you do not understand. If you choose not to participate in this data banking and data sharing study you will not be penalized or lose any benefits that you would otherwise be entitled to.

#### What will Happen to Your Genetic Data:

If you agree to this data banking and data sharing study, your genetic data and any other data that is collected in the study will be placed into a secure location(a large computer) at the University of Florida (UF). The results of your genetic tests will also go into your electronic medical record at Shands. Once the other study you agreed to (listed above) is completed, your genetic data and other data collected on you during that study will have all identifiable information removed and then be sent to the NIH data bank. Your deidentified data that is sent will be given a unique ID number, but only those at UF or your affiliated institution will be able to match this unique ID number to identify you.

IRB Project #: 201601774 
IRB Version: 10/19/2011



#### Who Can Use Your Stored Data:

At the NIH, de-identified genetic data that has been collected from you and other participants may be given to researcher from around the country who apply to the NIH to receive de-identified data to use in their research projects. This request will first have to be approved by an NIH committee that oversees the release of the data. Once the NIH committee approves the release of the de-identified data, the researcher will have to get local Institutional Review Board (IRB - an IRB is a group of people who are responsible for looking after the rights and welfare of people taking part in research) approval before they can start their study and use this de-identified genetic data

At the NIH, since your data is de-identified in the data bank, neither you nor UF nor your affiliated institution will receive any information when data is used in future research or receive any results from that future research.

#### **Benefits to You in Storing Your Data:**

There is no direct benefit to you for participating in this data bank.

#### **Risks to You in Storing Your Data:**

#### At NIH:

- Risk of Identification: The genetic data being sent to the NIH Data Bank is deidentified, however there is a slight chance that identifiable information may be mistakenly sent.
- Risk Associated with the Freedom of Information Act: Your information that is sent to the NIH will be kept in an NIH data bank and will, thereby, become U.S. government records that are subject to the Federal Freedom of Information Act (FOIA). As an agency of the Federal government, the NIH is required to release government records in response to requests under the federal Freedom of Information Act (FOIA), unless the records are exempt from release under one of the FOIA exemptions. The NIH believes that the only release of your data under such a request would be your data with the unique ID number removed.

IRB Project #: 201601774 
IRB Version: 10/19/2011

Study ID:IRB201601774 Date Approved: 10/18/2017 Expiration Date: 11/2/2018



• Risks Associated with Law Enforcement Access: It is possible that law enforcement agencies could request access to the de-identified genetic data within the NIH data bank and, for example, search for matches to DNA data collected as part of some criminal activity. While this is expected to be rare, such requests may be granted by the NIH. Law enforcement officials might then try to identify you by requiring your study doctor to release the key to the unique ID number which could identify you. However, the release of identifiable information by your study doctor may be protected by the Certificate of Confidentiality.

In order to better protect access to your genetic information, both UF and the NIH have obtained a Certificate of Confidentiality. Certificates of Confidentiality are issued by the National Institutes of Health (NIH) to protect researchers from being forced to release research records, which in this case is your genetic information. These Certificates allow the researchers and others who have access to research information to refuse to release information on research participants in any civil, criminal, administrative, legislative, or other proceeding, whether at the federal, state, or local level.

Risks to Specific Populations, Groups, and Communities: Medical research has
already shown that some populations demonstrate a higher likelihood to develop
certain medical diseases than others. It is possible that if you have some rare
condition or rare physical characteristics, that someone could identify you based
on the de-identified data in the NIH data bank.

#### Can You Withdraw Your Consent to Store Your Data?

If you decide that your genetic and clinical data can be kept for research but you later change your mind, tell the study staff listed in question #3 who will remove your data from the UF databank, and inform the Federal Data bank to remove your de-identified data from the data bank. There will be no cost to you for this storage of your de-identified genetic data.

#### Do You Agree to Participate?

Please review the statement below and <u>initial by your choice</u>:

I agree to have my de-identified genetic data shared with the NIH databank (dbGaP) to be used for future unknown research.

| Initials | YES | Initials | NO |
|----------|-----|----------|----|

IRB Project #: 201601774 IRB Version: 10/19/2011 PI Version: 11/21/2016